CLINICAL TRIAL: NCT04422938
Title: Mechanical Versus Manual Chest Compression: A Retrospective Study in In-hospital Cardiac Arrest
Brief Title: Mechanical Versus Manual Cardiopulmonary Resuscitation
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Alp Şener, Clinical Assistant Professor, Ankara City Hospital Bilkent
Other Study IDs: medybu-IN
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cardiac Arrest; Resuscitation
Keywords: Cardiopulmonary Resuscitation; Chest compression; In-hospital; Mechanical; Manuel
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Manuel compression: Manuel chest compressions will be handled by clinicians
  Interventions: Other: Manuel chest compressions handled by clinicians
- Mechanical compression: Mechanical chest compressions will be handled via mechanical chest compression device
  Interventions: Device: LUCAS™ 2 Chest Compression System

INTERVENTIONS:
Other: Manuel chest compressions handled by clinicians — Compressions will be handled by human efforts
  Groups: Manuel compression
Device: LUCAS™ 2 Chest Compression System — LUCAS-2 model piston-based mechanical chest compression device was used for mechanical chest compressions
  Groups: Mechanical compression

SUMMARY:
In this study, the investigators compared mechanical and manual chest compressions in in-hospital cardiac arrest cases.

DETAILED DESCRIPTION:
In this study, the investigators analyzed cardiopulmonary resuscitations performed over a 2-year period in an emergency department of a training and research hospital and compared success of manual and mechanical chest compressions in terms of return of spontaneous circulation, 30-day survival, and hospital discharge. Investigators present the study as an in-hospital cardiac arrest study; however, all of the resuscitation performed in the cases included in the study were performed in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

Over 18 age Cardiac arrest cases In-hospital cardiac arrest cases Resuscitations performed in emergency department

Exclusion Criteria:

<18 age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with cardiac arrest in-hospital environment (in emergency department) and whose had manual or mechanical cardiopulmonary resuscitation in emergency department included in the study; data were collected hospital management information system and analyzed retropectively.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate on the 30th day | 30 days
  Mortality rates from the hospital admission to the 30th day
Rate of the return of spontaneous circulation | 5 minutes
  Rate of return of the spontaneous circulation with duration at least five minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, School of Medicine, Department of Emergency Medicine, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.

REFERENCES:
- [Background] Couper K, Yeung J, Nicholson T, Quinn T, Lall R, Perkins GD. Mechanical chest compression devices at in-hospital cardiac arrest: A systematic review and meta-analysis. Resuscitation. 2016 Jun;103:24-31. doi: 10.1016/j.resuscitation.2016.03.004. Epub 2016 Mar 11. PMID 26976675
- [Background] Couper K, Quinn T, Lall R, Devrell A, Orriss B, Seers K, Yeung J, Perkins GD; COMPRESS-RCT collaborators. Mechanical versus manual chest compressions in the treatment of in-hospital cardiac arrest patients in a non-shockable rhythm: a randomised controlled feasibility trial (COMPRESS-RCT). Scand J Trauma Resusc Emerg Med. 2018 Aug 30;26(1):70. doi: 10.1186/s13049-018-0538-6. PMID 30165909